CLINICAL TRIAL: NCT01422746
Title: Effect of Metformin on Adrenal or Ovarian Androgen Production in Overweight Pubertal Girls With Androgen Excess (CBS005)
Brief Title: Effect of Metformin on Adrenal or Ovarian Androgen Production in Overweight Pubertal Girls With Androgen Excess
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19302; CBS006 (Other: University of Virginia)
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Hyperandrogenemia; Polycystic Ovary Syndrome
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- metformin (Experimental): 12 weeks metformin, with pre- and post- dexamethasone and ACTH to perform standardized adrenal stimulation testing; dexamethasone and rhCG to perform standardized ovarian stimulation testing
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500-1000 mg PO BID (X12 weeks)
  Other Names: Glucophage

SUMMARY:
This study will test whether metformin administration can ameliorate androgen (male hormone) overproduction in overweight pubertal girls with androgen excess. The investigators hypothesize that improvement in insulin sensitivity by 12 weeks of metformin administration will improve androgen levels after adrenal stimulation testing with adrenocorticotropic hormone (ACTH) or ovarian stimulation testing with recombinant human chorionic gonadotropin (rhCG).

ELIGIBILITY:
Inclusion Criteria:

* Overweight(>85th BMI%) females
* Early to late puberty (expected age range 7-18)
* Hyperandrogenemic (free testosterone greater than 2.5 standard deviations above the mean for normal control subjects of the same Tanner Stage)
* Screening labs within age-appropriate normal range, with the exception of a mildly low hematocrit (see below) and the hormonal abnormalities inherent in obesity which could include mildly elevated luteinizing hormone (LH), lipids, testosterone, prolactin, DHEAS, E2, glucose, and insulin; and decreased follicle-stimulating hormone (FSH) and/or sex hormone-binding globulin (SHBG)

Exclusion Criteria:

* Age < 7 or > 18 y
* Inability to comprehend what will be done during the study or why it will be done
* BMI-for-age < 5th percentile
* Positive pregnancy test or lactation.
* Abnormal laboratory studies will be confirmed by repeat testing to exclude laboratory error.
* Morning cortisol < 3 µg/dL or history of Cushing syndrome or adrenal insufficiency
* History of congenital adrenal hyperplasia or 17-hydroxyprogesterone > 300 ng/dL, which suggests the possibility of congenital adrenal hyperplasia (if postmenarcheal, the 17-hydroxyprogesterone will be collected during the follicular phase, or ≥ 40 days since last menses if oligomenorrheic). NOTE: If a 17-hydroxyprogesterone >300 mg/dL is confirmed on repeat testing, an ACTH-stimulated 17-hydroxyprogesterone <1000 ng/dL will be required for study participation.
* Total testosterone > 150 ng/dL, which suggests the possibility of a virilizing neoplasm
* DHEAS greater than the upper limit of age-appropriate normal range (mild elevations may be seen in polycystic ovary syndrome (PCOS) and adolescent hyperandrogenemia (HA), and elevations < 1.5 times the age-appropriate upper limit of normal will be accepted in these groups)
* Virilization
* Previous diagnosis of diabetes, fasting glucose ≥126 mg/dL, or a hemoglobin A1c ≥6.5%
* Abnormal thyroid stimulating hormone (TSH) for age. Subjects with stable and adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded.
* Abnormal prolactin. Mild elevations may be seen in overweight girls, and elevations <1.5 times the upper limit of normal will be accepted in this group.
* Persistent hematocrit <36% and hemoglobin <12 g/dL. Subjects with a mildly low hematocrit (33-36%) will be asked to take iron in the form of ferrous gluconate for up to 60 days. Subjects weighing ≤ 36 kg will take one 300-325 mg tablet oral ferrous gluconate daily (containing 36 mg elemental iron);subjects weighing >36 kg will take two 300-325 mg tablets oral ferrous gluconate daily (containing 36 mg elemental iron each). They will return to the Clinical Research Unit (CRU) after 30-60 days of iron therapy to have their hemoglobin or hematocrit rechecked and will proceed with the remainder of the study if it is ≥12 g/dL or ≥36%, respectively.
* Persistent liver test abnormalities, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Mild elevations may be seen in overweight girls, so elevations <1.5 times the upper limit of normal will be accepted in this group.
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Abnormal sodium, potassium, or bicarbonate concentrations, or elevated creatinine concentration (confirmed on repeat)
* No medications known to affect the reproductive system or glucose metabolism can be taken in the 3 months prior to the study. Such medications include oral contraceptive pills, progestins, metformin, glucocorticoids, and psychotropics.

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in free testosterone or 17-hydroxyprogesterone levels after ACTH and rhCG administration respectively, before and after metformin administration for 12 weeks | 12 weeks after metformin administration

SECONDARY OUTCOMES:
Changes in adrenal and ovarian steroid precursors after ACTH and rhCG; body composition via air displacement plethysmography, BMI, and glucose tolerance testing results; baseline and after 12 weeks of metformin administration | 12 weeks after metformin administration

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No